CLINICAL TRIAL: NCT02310997
Title: Transplantation Of Umbilical Cord Blood From Unrelated Donors In Patients With Haematological Diseases Using A Myeloablative Conditioning Regimen
Brief Title: Myloablative Cord Blood Transplant in Haematological Malignancies (MAC UCBT)
Acronym: MAC UCBT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial closed early due to poor recruitment
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/09/0128; 2009-011818-21 (EudraCT Number)
Record Dates: First submitted 2014-09-18; First posted 2014-12-08 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Leukaemia; Lymphoma; Other Haematological Diseases
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — Cyclophosphamide; Whole-Body Irradiation; Busulfan; Melphalan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fludarabine + Cyclophosphamide + TBI (Experimental): Patients aged 2-45 years (excluding AML, JMML and MDS patients aged <16 years) will receive an umbilical cord blood transplant using a myeloablative conditioning regimen comprising:
  Fludarabine 25mg/m^2/day day -8 to -6 (total 75mg/m^2) Cyclophosphamide 60mg/kg day -7 and -6 (total 120mg/kg) Total body irradiation 13 - 14.4Gy in 6-8 fractions
  Interventions: Other: Umbilical Cord Blood Transplant; Drug: Cyclophosphamide; Radiation: Total body irradiation; Drug: Fludarabine
- Busulfan + Cyclophosphamide + Melphalan (Experimental): Patients aged < 2 years and AML, JMML and MDS patients <16 years will receive an umbilical cord blood transplant using a myeloablative conditioning regimen comprising:
  Busulfan 3.2mg/kg/day in 2 or 4 doses per day, days -9 to -6 (total 12.8mg/kg). Cyclophosphamide 60mg/kg days -4 and -3 (total 120mg/kg) Melphalan 140mg/m^2 day -2
  Interventions: Other: Umbilical Cord Blood Transplant; Drug: Cyclophosphamide; Drug: Busulfan; Drug: Melphalan

INTERVENTIONS:
Other: Umbilical Cord Blood Transplant
Drug: Cyclophosphamide
Radiation: Total body irradiation
  Arms: Fludarabine + Cyclophosphamide + TBI
Drug: Busulfan
  Arms: Busulfan + Cyclophosphamide + Melphalan
Drug: Melphalan
  Arms: Busulfan + Cyclophosphamide + Melphalan
Drug: Fludarabine
  Arms: Fludarabine + Cyclophosphamide + TBI

SUMMARY:
This trial is looking at using umbilical cord blood from unrelated donors after high dose chemotherapy. It is for people who have cancer of the bone marrow or lymphatic system including leukaemia and lymphoma, or a blood disorder called myelodysplastic syndrome (MDS).

The trial is for babies over 4 weeks old, children, and adults up to the age of 45.

DETAILED DESCRIPTION:
During treatment for cancers of the bone marrow or lymphatic system, a lot of the stem cells are damaged and you may need a bone marrow or stem cell transplant to replace them.

Stem cells can also be collected from the umbilical cord of newborn babies. Many people around the world have donated their baby's umbilical cords which are stored safely.

There are usually enough cells in one cord to transplant a small child, but there may not be enough cells for an older child or adult. Researchers want to see if adults and children can safely have stem cells from more than 1 umbilical cord.

Before a transplant, you have high doses of chemotherapy, sometimes with radiotherapy. This intensive conditioning aims to destroy all the cells in your bone marrow, and is called myeloablative conditioning.

The aim of this trial is to see if a transplant using cord blood cells from unrelated donors after myeloablative conditioning is safe, and whether it helps people who need a stem cell transplant but don't have a stem cell donor.

You may be able to enter this trial if you:

* Have leukaemia, lymphoma or another disorder of the bone marrow and treatment with intensive conditioning followed by a stem cell transplant is likely to help you
* Do not have a suitable stem cell donor in your family, and your doctors have not been able to find a matched unrelated donor
* Have satisfactory blood test results
* Are between 4 weeks and 45 years old

You cannot enter this trial if you:

* Have a family member who could donate stem cells to you, or you have a matched unrelated donor
* Can have any other treatment that your doctors think will cure your disease or keep it under control for a long time
* Have already had a lot of radiotherapy (the trial doctor can advise you about this)
* Have already had a bone marrow or stem cell transplant using your own cells
* Have chronic myeloid leukaemia that is in chronic phase and is responding to imatinib, or is in blast phase and is not responding to treatment Have acute lymphoblastic leukaemia that is not responding to treatment or has come back and more than 5% of your bone marrow is made up of immature cells (blasts)
* Have acute myeloid leukaemia that is not responding to treatment or has come back and more than 20% of your bone marrow is made up of immature cells (blasts)
* Have a disease that has come back and you are having another type of treatment (salvage treatment) but your disease is not responding or is getting worse
* Have a blood disorder called myelofibrosis
* Have a blood disorder called aplastic anaemia
* Have an infection that cannot be controlled with medication
* Have either the HIV or HTLV virus
* Are pregnant or breastfeeding

This phase 2 trial aims to recruit 60 people. It will include both adults and children. Everybody taking part will have intensive conditioning before having a transplant of stem cells from the umbilical cord blood of at least 1 unrelated donor.

To take part in this trial, the researchers need to be sure that there are 2 lots of cord blood cells that would be suitable for you. They will only use cells from 2 cords if there is some concern that they won't get enough cells from 1 umbilical cord.

People aged between 2 and 45 (apart from children under the age of 16 who have acute myeloid leukaemia, juvenile myelomonocytic leukaemia (JMML) or MDS) will have conditioning with fludarabine, cyclophosphamide and radiotherapy to the whole body (total body irradiation). This takes 9 days all together. On the last day, you have the stem cells through a drip into a vein.

Children under 2 years of age (and children up to the age of 16 who have acute myeloid leukaemia, JMML or MDS) will have conditioning with busulfan, cyclophosphamide and melphalan. They do not have radiotherapy. This conditioning takes 10 days all together. They have the stem cells through a drip into a vein on the 11th day.

The stem cells find their way into your bone marrow where they will start making new blood cells.

You will see the trial team and have some tests before you start treatment. The tests include:

* Physical examination
* Blood tests
* Chest X-ray
* Lung function tests
* Heart trace (ECG)
* Heart ultrasound (echocardiogram) or MUGA scan
* Bone marrow test When you have your treatment, you will be in hospital for about 4 to 6 weeks. As you will be at a high risk of infection, you will be in your own room. This is called being in isolation. You have another bone marrow test a month after your transplant.

When you go home, you have to go back to the hospital for regular blood tests. This is likely to be 2 or 3 times a week to begin with. You may have to go back into hospital for a few days at some point.

After a transplant, you will see the doctors and have blood tests At least once a week for the first 3 months At least once a month for the rest of the first year The trial doctors will follow your progress closely for at least 2 years.

The main side effect of the treatment you have just before the transplant is a drop in the number of blood cells, causing an increased risk of infection, tiredness and breathing problems.

We have more information about fludarabine, cyclophosphamide, busulfan and melphalan in our cancer drugs section.

It takes longer for blood cells to start growing again after a transplant of cord blood than after other types of stem cell transplant. Even when your blood count gets back to normal, your immune system may take up to 2 years to recover fully.

Unfortunately, this treatment can affect your ability to have children (your fertility). Men taking part will be offered the option to store sperm (sperm banking) before starting treatment. Preserving fertility for women is more complicated and it is important that women talk to their doctors about this before starting treatment.

After any type of bone marrow or stem cell transplant, there is a risk of graft versus host disease (GVHD). This happens when the new stem cells attack your body tissue. It mainly affects your skin, gut and liver.

Rarely, the new stem cells fail to start working. This is more common with cord blood transplants than with other bone marrow transplants. And even if your transplant is successful, there is a risk your disease may come back. Because of these risks, your doctors will monitor you very closely after your transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be < 45 years of age and ≥ 28 days old
* Patients with high risk, advanced or poorly responding haematological disease for which there is published evidence that haematopoietic stem cell transplantation using myeloablative conditioning is likely to be effective
* The individual patient's disease status is such that there is no alternative therapy likely to achieve cure or provide a significant prolongation of disease-free survival
* Left ventricular ejection fraction >45%
* Transaminases and bilirubin < twice the upper limit of the normal range
* Creatinine clearance > 60mls/min
* Comorbidity index of 0 or 1

Exclusion Criteria:

* Patients with a suitably matched sibling donor or 10/10 unrelated volunteer donor available within an acceptable time period.
* Pregnancy or breastfeeding.
* Evidence of HIV or HTLV (I+II) infection or known HIV or HTLV positive serology
* Current active serious infection, in particular uncontrolled fungal infection -Previous irradiation that precludes the safe administration of an additional dose of 13- 14.4 Gy of total body irradiation (TBI) in patients aged 2-45 years
* Prior autograft
* CML in first chronic phase responding to Imatinib or refractory blast crisis
* Patients with acute leukaemia in morphological relapse/ persistent disease (defined as > 5% blasts in normocellular bone marrow)
* Patients with acute myeloid leukaemia with relapse/persistent disease unresponsive to re-induction chemotherapy (defined as >20% blasts in normocellular bone marrow)
* Malignant disease that is refractory to or progressive on salvage therapy
* Myelofibrosis.
* Aplastic anaemia

Ages: 28 Days to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Non-relapse mortality at 100 days post transplant | 100 days post transplant

SECONDARY OUTCOMES:
Overall survival at 1 year | 1 year post transplant
Time course of mixed chimerism established by the donor graft | 28, 60, 100 days, 6 months, 1 year post transplant
Recovery from neutropenia and cytopenia | up to 1 year post transplant
Incidence of acute and chronic GVHD | 100 Days and 1 year post transplant
Incidence of relapse | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Hough, Principal Investigator — University College London Hospital
Locations (12):
- United Kingdom (12):
  - University College London Hospital, London, Greater London
  - University Hospital Birmingham, Birmingham
  - Bristol Haematology & Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - St James' University Hospital, Leeds
  - St Bartholomew's Hospital, London
  - Great Ormond Street Hospital for Children, London
  - Manchester Royal Infirmary, Manchester
  - Christie Hospital NHS Foundation Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Royal Hallamshire Hospital, Sheffield
  - Royal Marsden Hospital, Sutton